CLINICAL TRIAL: NCT02739438
Title: The Study of ELEctronic Cigarette Toxicity in a Human Model in Vivo Model of Inflammation and Vascular Dysfunction (SELECT)
Brief Title: The Study of ELEctronic Cigarette Toxicity in a Human Model in Vivo Model of Inflammation and Vascular Dysfunction
Acronym: SELECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Murali Shyamsundar, Senior lecturer and Consultant in Intensive Care Medicine, Queen's University, Belfast
Other Study IDs: B16/28
Record Dates: First submitted 2016-04-11; First posted 2016-04-15 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Acute Lung Injury
Keywords: Pulmonary inflammation; Endothelial dysfunction; Electronic Cigarettes
MeSH Terms: conditions — Acute Lung Injury; Pneumonia; Vaping | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken at initially for screening then at baseline, 24 hours after first bronchoscopy, prior to the inhalation of LPS 6 weeks later and 24 hours post LPS inhalation.
  Urine sample will be collected before both camera tests. Bronchoalveolar lavage fluid will be taken at baseline then 6 weeks later.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- E Cigarette users: Subjects who use electronic cigarettes daily and have not used conventional cigarettes in the previous 3 months. Total pack years of smoking should be less than 20 for their smoking history, with normal lung function (FEV1 and FEV1/FVC) and no clinical symptoms of airway obstruction/inflammation (cough, dyspnea, sputum and wheeze).
  Interventions: Other: Electronic cigarette use
- Cigarette smokers: Subjects who smoke at least ¼ pack cigarettes per day for the past 1 year, with no history of electronic cigarette use in the last 30 days.
  Interventions: Other: Cigarette use
- Control group: Subjects with no history of prior conventional cigarette (< 100 cigarettes lifetime) or electronic cigarette use.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Electronic cigarette use — Subjects who use electronic cigarettes daily and have not used conventional cigarettes in the previous 3 months.
  Groups: E Cigarette users
Other: Cigarette use — Subjects who smoke at least ¼ pack cigarettes per day for the past 1 year, with no history of electronic cigarette use in the last 30 days.
  Groups: Cigarette smokers
Other: Control group — Subjects with no history of prior conventional cigarette (< 100 cigarettes lifetime) or electronic cigarette use.
  Groups: Control group

SUMMARY:
To carry out a prospective cohort study of healthy volunteers, assessing differences between baseline pulmonary inflammation, response to LPS inhalation and endothelial function, as measured by flow mediated dilation between, electronic cigarette uses, cigarette smokers and non smokers.

DETAILED DESCRIPTION:
Background. Since their introduction, electronic cigarette (EC) use has increased substantially. Perhaps most concerning is the increased use amongst adolescents. Many e-cigarette users believe that electronic cigarettes are safer than conventional cigarettes [1]. However, the toxicities of electronic cigarettes, including those in the lung, are relatively poorly studied. Notably, early studies suggest that electronic cigarettes are not harmless. The fine and ultra-fine particles could deposit in the lungs and lead to harm. Animal studies of electronic cigarettes have been associated with a number of pulmonary toxicities, including increased inflammation and oxidative stress in the lung [2] as well as impaired pulmonary immunity [3, 4]. EC vapour reduces indoor air quality by increasing the concentrations of particulate matter, particle number concentrations, polycyclic aromatic hydrocarbons (PAH) which are known carcinogens [5]. Early studies on cardiovascular function also suggests harm from the constituents of EC vapour such as the direct effects of nicotine, carbonyls as well as fine and ultrafine particles [6].

There is limited understanding of the adverse effects of EC vapour of the pulmonary or cardiovascular physiology and additional studies, particularly in humans, are needed to better characterize the acute toxicities of electronic cigarettes

Hypothesis Our hypothesis is, when compared to cigarette or e-cigarette naïve healthy volunteers;

1. E-cigarette users will have a higher baseline pulmonary inflammation
2. E-cigarette users will have an exaggerated immune response after LPS inhalation
3. E-cigarettes users will have endothelial dysfunction as measured by FMD of the brachial artery

Trial design Prospective cohort study of healthy subjects exposed to inhaled LPS.

Population Healthy subjects, including electronic cigarette users, cigarette smokers and controls will be recruited by advertising.

Intervention Bronchoscopy and blood sampling to assess baseline pulmonary and systemic inflammation and injury and in response to inhaled LPS 50 mcg. Flow mediated dilation (FMD) of brachial artery to study endothelial dysfunction.

After informed consent, their baseline FMD of brachial artery will be measured as well as lung function. FMD of brachial artery will be measured within 5 mins of use of e-cigarette to reflect the acute effects of e-cigarette on systemic endothelial dysfunction. Bronchoscopy with BAL, blood and urine sampling will be performed. This will enable us to measure the baseline inflammation and markers of cellular injury without inhaled LPS. At 24 hours the subject will return and lung function will be measured and blood sampling will be performed.

Six weeks later, the above procedure will be repeated but with LPS stimulation. The subject will once again attend the hospital and lung function will be measured, blood and urine sampling will be performed. Subjects will inhale LPS (from Escherichia coli O26:B6, 50 μg; Sigma-Aldrich, St. Louis, MO) using a dosimeter. Bronchoscopy with BAL will be undertaken 6 hours following LPS inhalation. Prior to bronchoscopy, lung function will be measured in order to ensure that they may safely undergo LPS inhalation. At 24 hours subjects will return and lung function will be measured and blood sampling will be performed. The time points for BAL and plasma sampling are chosen to obtain insight into both cytokine/chemokine release and neutrophil recruitment after pulmonary delivery of LPS.

Statistical considerations The primary exposure variable will be e-cigarette exposure; the primary outcome variable will be plasma and BAL biomarkers of injury and inflammation. Given that early studies of electronic cigarettes suggest that they may be associated with inflammation, we have used BAL absolute neutrophil count, a key marker of inflammation, to inform our sample size. Based on data from controls in our prior study, a cohort of 10 e-cigarette users and 10 controls should be able to detect a minimal difference of 7.09 x 105 cells in the BAL after LPS inhalation between groups with 80% power using Wilcoxon Rank Sum testing. Of note, this is similar to the difference we observed between smokers and non-smokers after LPS in our prior study [7]. Additionally, we will compare biomarkers of inflammation and injury in electronic cigarette users to those from conventional cigarette smokers using Wilcoxon Rank Sum testing. All data will be analysed using STATA 13.1 (StataCorp LP, College Station, TX).

Study Monitoring Site monitoring will be directed by the sponsor according to the study risk assessment. Site visits will be performed on a regular basis as required by the sponsor to ensure that all regulatory requirements are met and to monitor the quality of the data collected. The CRF will be used for source data verification.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects less than 45 years of age and BMI < 35

Exclusion Criteria:

1. Age < 18 years
2. Pregnant or Breast-Feeding
3. Participation in a clinical trial of an investigational medicinal product within 30 days
4. Consent declined
5. History of asthma
6. Marijuana use or other inhaled products with or without nicotine in the last 3 months
7. Alcohol abuse, as defined by the Alcohol Use Disorders Identification Test (AUDIT)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects, including electronic cigarette users, cigarette smokers and controls will be recruited.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
bronchoalveolar lavage neutrophil count in response to LPS stimulation | BAL 6 hours after LPS inhalation

SECONDARY OUTCOMES:
Alveolar inflammatory response | 24 hours after LPS inhalation
  1. Alveolar inflammatory response biomarkers which may include but are not limited to the measurement of BAL cytokines (including but not limited to TNFα, IL1β, IL6, IL8), proteases and antiproteases, HO1, coagulation factors (including but not limited to thrombin-antithrombin complex, tissue factor, protein C, thrombomodulin and plasminogen activator inhibitor1), and RAGE ligands. Identification of specific cellular populations within the BAL (using but not limited to cytospins, flow cytometry, ELISpot assays, in vitro cell expansion).
Plasma inflammatory response | 24 hours after LPS inhalation
  Plasma inflammatory response biomarkers which may include but are not limited to measurement of plasma CRP, cytokines (including but not limited to TNFα, IL1β, IL6, IL8), proteases and antiproteases, HO1, adhesion and activation molecule expression (including but not limited to sICAM1), coagulation factors (including but not limited to thrombin-antithrombin complex, tissue factor, protein C, thrombomodulin and plasminogen activator inhibitor1), and RAGE ligands.
Indices of alveolar epithelial and endothelial and injury | 24 hours after LPS inhalation
  Intracellular signalling activity in the alveolar space which may include but not limited to the measurement of BAL total and phosphorylated p38, ERK and JNK MAPKs and STAT -1/-3 from leucocyte extracts. Activated and total IκBα and β will be measured in cytoplasmic extracts and NFκβ and AP-1 in nuclear extracts.
4. FMD of brachial artery as a marker of the effects of e-cigarettes on endothelial function | 5 mins within use of an electronic cigarette
  FMD of brachial artery to study endothelial dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Murali Shyamsundar, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queens University, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutten LJ, Blake KD, Agunwamba AA, Grana RA, Wilson PM, Ebbert JO, Okamoto J, Leischow SJ. Use of E-Cigarettes Among Current Smokers: Associations Among Reasons for Use, Quit Intentions, and Current Tobacco Use. Nicotine Tob Res. 2015 Oct;17(10):1228-34. doi: 10.1093/ntr/ntv003. Epub 2015 Jan 14. PMID 25589678
- [Background] Lerner CA, Sundar IK, Yao H, Gerloff J, Ossip DJ, McIntosh S, Robinson R, Rahman I. Vapors produced by electronic cigarettes and e-juices with flavorings induce toxicity, oxidative stress, and inflammatory response in lung epithelial cells and in mouse lung. PLoS One. 2015 Feb 6;10(2):e0116732. doi: 10.1371/journal.pone.0116732. eCollection 2015. PMID 25658421
- [Background] Wu Q, Jiang D, Minor M, Chu HW. Electronic cigarette liquid increases inflammation and virus infection in primary human airway epithelial cells. PLoS One. 2014 Sep 22;9(9):e108342. doi: 10.1371/journal.pone.0108342. eCollection 2014. PMID 25244293
- [Background] Sussan TE, Gajghate S, Thimmulappa RK, Ma J, Kim JH, Sudini K, Consolini N, Cormier SA, Lomnicki S, Hasan F, Pekosz A, Biswal S. Exposure to electronic cigarettes impairs pulmonary anti-bacterial and anti-viral defenses in a mouse model. PLoS One. 2015 Feb 4;10(2):e0116861. doi: 10.1371/journal.pone.0116861. eCollection 2015. PMID 25651083
- [Background] Schober W, Szendrei K, Matzen W, Osiander-Fuchs H, Heitmann D, Schettgen T, Jorres RA, Fromme H. Use of electronic cigarettes (e-cigarettes) impairs indoor air quality and increases FeNO levels of e-cigarette consumers. Int J Hyg Environ Health. 2014 Jul;217(6):628-37. doi: 10.1016/j.ijheh.2013.11.003. Epub 2013 Dec 6. PMID 24373737
- [Background] Morris PB, Ference BA, Jahangir E, Feldman DN, Ryan JJ, Bahrami H, El-Chami MF, Bhakta S, Winchester DE, Al-Mallah MH, Sanchez Shields M, Deedwania P, Mehta LS, Phan BA, Benowitz NL. Cardiovascular Effects of Exposure to Cigarette Smoke and Electronic Cigarettes: Clinical Perspectives From the Prevention of Cardiovascular Disease Section Leadership Council and Early Career Councils of the American College of Cardiology. J Am Coll Cardiol. 2015 Sep 22;66(12):1378-91. doi: 10.1016/j.jacc.2015.07.037. PMID 26383726